CLINICAL TRIAL: NCT03347305
Title: Study in Calorimetric Room of the Energy Metabolism of Renal Impairment Patients Treated With Automated Peritoneal Dialysis
Brief Title: Measurement of the Energy Metabolism of Peritoneal Dialysis Patients
Acronym: CALIMERO 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Pôle Santé République (Other); Service de Néphrologie et Hémodialyse (Unknown); Jacques Lacarin Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-364; 2015-A00035-44 (Other: 2015-A00035-44)
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Renal Failure
Keywords: Energy expenditure; Peritoneal dialysis
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Group DPA (Experimental): The main objective is to compare DE and its variations according to the conditions (rest, sleep, meals, physical activity) in patients treated with automated DP compared to controls, in a calorimetric chamber
  Interventions: Behavioral: automated DP
- Healthy Volunteers (Experimental): The main objective is to compare DE and its variations according to the conditions (rest, sleep, meals, physical activity) in patients treated with automated DP compared to controls, in a calorimetric chamber
  Interventions: Behavioral: Calorimetric chamber

INTERVENTIONS:
Behavioral: automated DP — Energy expenditure measurement
  Arms: Patients Group DPA
Behavioral: Calorimetric chamber — The main objective is to compare DE and its variations according to the conditions (rest, sleep, meals, physical activity) in patients treated with automated DP compared to controls, in a calorimetric chamber
  Arms: Healthy Volunteers

SUMMARY:
The daily energy expenditure of patients treated with peritoneal dialysis could be increased compared to the general population and promote the development of a state of undernutrition. Conversely, the absorption of glucose by transperitoneal route could contribute to the occurrence of a metabolic syndrome.

The main objective is to compare DE and its variations according to the conditions (rest, sleep, meals, physical activity) in patients treated with automated DP compared to controls, in a calorimetric chamber.

DETAILED DESCRIPTION:
The daily energy expenditure of patients treated with peritoneal dialysis could be increased compared to the general population and promote the development of a state of undernutrition. Conversely, the absorption of glucose by transperitoneal route could contribute to the occurrence of a metabolic syndrome.

The main objective is to compare DE and its variations according to the conditions (rest, sleep, meals, physical activity) in patients treated with automated DP compared to controls, in a calorimetric chamber.

ELIGIBILITY:
Inclusion Criteria:

* Patients Group DPA

  * Male patients
  * Aged 18 to 70 years
  * With end-stage renal disease
  * Treated by automatic peritoneal
  * Social security cover
  * Without acute events in the 3 months prior to inclusion
  * PCR < 30 mg/L
  * Written informed consent
  * Baecke activity score from 5 to 10

Healthy Volunteers

* Male patients
* Aged 18 to 70 years
* Patients matched by lean body mass (± 2 kgs) and age (± 5 years)
* Having a glomerular filtration rate estimated with the formula CKD-EPI creatinine > 60 mL / min / 1.73 m 2
* PCR < 3 mg/L
* Social security cover
* Written informed consent
* Baecke activity score from 5 to 10

Exclusion Criteria:

* • - Female

  * Type 1 or 2 diabetes requiring a antidiabetic treatment
  * Decompensated heart failure
  * Smoking more than 5 cigarettes a day
  * Alcoholic patients, drinking more than 3 glass of alcohol a day
  * Patient Corticotherapy in progress
  * Patient with evolutive acute pathology
  * Person who has participated in another study within the last 30 days or is in period of exclusion on the National File of Healthy Volunteers

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure measured by indirect calorimetry in a calorimetric chamber | at day 1
  Energy expenditure measured by indirect calorimetry in a calorimetric chamber

SECONDARY OUTCOMES:
respiratory quotient (RQ) | at day1
  Nature of the oxidized nutrients determined from the measurement of the respiratory quotient
Actimetry | at day 1
  Estimated ambulatory energy expenditure from heart rate
HGPO | at day 1
  Charges of blood insulin concentration, and glucose in response to oral glucose load

CONTACTS AND LOCATIONS:
Overall Officials: Julien ANIORT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France